CLINICAL TRIAL: NCT00466674
Title: Treatment of Myeloma in Patients <= 65 Years Old With Response >= 50% After HSC Autotransplant by Allogenic Transplant Genoidentical or Phenoidentical After Reduced Intensity Conditioning (IFM 2005-03)
Brief Title: Treatment of Myeloma in Patients <= 65 Years Old With Response >= 50% After HSC Autotransplant by Allogenic Transplant Genoidentical or Phenoidentical After Reduced Intensity Conditioning
Acronym: IFM 2005-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005.385
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myeloma
Keywords: Myeloma; RICT; conditioning; allograft
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogenic Transplant (Experimental)
  Interventions: Drug: reduced intensity conditioning

INTERVENTIONS:
Drug: reduced intensity conditioning — reduced intensity conditioning for allogenic transplant

SUMMARY:
Donor mobilization :

Donor will be mobilized with G-CSF (Granocyte) sub-cutaneous 10 µg/kg/day during 5 to 6 days.

Hematopoïetic Stem Cell Harvest:

By 1, 2, or 3 aphaeresis, a number of 4 x 106 cellules CD34+ /kg is required. If the CD34+ >= 2 and <= 4x106/kg: the center must decide on the strategy Decision. In case of insufficient graft : a Bone Marrow Harvest is recommended Conditioning : Fludarabine - Busulfan - ATG

* D-5 : Fludarabine (30 mg/m²)
* D-4 : Fludarabine (30 mg/m²)+ Busilvex (0,8 mg/kg every 6 h)
* D-3 : Fludarabine (30 mg/m²)+ Busilvex (0,8 mg/kg every 6 h)
* D-2 : Fludarabine (30 mg/m²) + ATG (Genzyme) (2.5 mg/Kg)
* D-1 : Fludarabine (30 mg/m²) + ATG (Genzyme) (2.5 mg/Kg) GVHD Prophylaxis: CsA alone at 3 mg/ kg + Methotrexate D1, D3 and D6 only in case of minor ABO incompatibility and with an anti A/B antibodies titer> 1/32.

Transplant : HSC at D0

• 3 months after Transplantation :

Disease Evaluation :

* If CR : Supervision. Then if progression: 4 cycles of Bortezomib.
* If no CR : Bortezomib (4 cycles)

  • Evaluation after Bortezomib cycles
* If CR : Supervision. Then, if progression and no GvHD : DLI If no RC and no GVHD : DLI

ELIGIBILITY:
Inclusion Criteria:

* Major patients not under guardianship
* Myeloma with high b2 microglobulin level (> 3 mg/l) and/or chromosome 13 deletion, and/or translocation t(4;14) stage I DS with high evolutive potential or stage II, III DS.

AND

* With response >= 50% and <= 90% after the first AutoHSCT (IFM 2005 01). The evaluation must be performed within 2 months after the first AutoHSCT.
* with an HLA identical related or unrelated donor ( match 10/10).
* Donor and recipient must have signed a written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Improvement of 15% of Event-free survival (EFS) at 3 years after allo HSCT (decrease of the number of deaths and progressions). | 3 years

SECONDARY OUTCOMES:
Haematological recovery | 3 years
Engraftment rate and graft failure rate | 3 years
The tolerance of Bortezomib after AlloHCST | 5 years
CR (Complete Response) length rate defined by Bladé criteria. | 5 years
Incidence and severity of acute and chronic GVHD | 5 years
Outcome of GVHD under treatment by Bortezomib | 5 years
Chimerism study by competitive PRC | 5 years
Immunological study of the graft (ancillary study) | 5 years
Study of immunological recovery by the recipient | 5 years
TRM = Transplant- Related Mortality at 3 months | 3 months
TRM = Transplant- Related Mortality at 1 year | 1 year
Study of quality of life | 5 years
Global survival at 3 years and 5 years | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette Michallet, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Mohamad Sobh, Lyon, France

REFERENCES:
- [Result] Michallet M, Sobh M, El-Cheikh J, Morisset S, Sirvent A, Reman O, Cornillon J, Tabrizi R, Milpied N, Harousseau JL, Labussiere H, Nicolini FE, Attal M, Moreau P, Mohty M, Blaise D, Avet-Loiseau H. Evolving strategies with immunomodulating drugs and tandem autologous/allogeneic hematopoietic stem cell transplantation in first line high risk multiple myeloma patients. Exp Hematol. 2013 Dec;41(12):1008-15. doi: 10.1016/j.exphem.2013.08.003. Epub 2013 Aug 29. PMID 23994781